CLINICAL TRIAL: NCT00002948
Title: A Phase I Study of High Dose Topotecan With Filgrastim and Peripheral Blood Stem Cell Support for Patients With Refractory Malignancies
Brief Title: High-Dose Topotecan and Peripheral Stem Cell Transplantation in Treating Patients With Refractory Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065416; YALE-HIC-9042; NCI-G97-1155
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Filgrastim; Topotecan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: topotecan hydrochloride
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of high-dose topotecan and peripheral stem cell transplantation in treating patients with refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, toxicities, and preliminary antitumor activity of escalating doses of topotecan, with filgrastim (G-CSF) and peripheral blood stem cell support, when administered to patients with refractory malignancies for which no effective therapy exists.

OUTLINE: This is a dose-escalation study.

Prior to stem cell harvesting, patients receive 1-2 courses of mobilizing salvage chemotherapy.

After stem cell harvest, high-dose topotecan is administered according to an escalating dosage scale. Topotecan is given over 30 minutes daily for three days. A minimum of 3 patients are entered at each dose level. The MTD is defined as the dose immediately below that at which 2 patients experience dose limiting toxicity.

Peripheral blood stem cells (PBSC) are infused at least 24 hours after treatment with topotecan is complete. Filgrastim (G-CSF) is administered subcutaneously beginning on the day PBSC are infused and continuing until blood counts recover.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed refractory malignancies for which no effective therapy is currently available

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3

Hepatic:

* Total bilirubin no greater than 2.0 mg/dL
* No chronic active hepatitis

Renal:

* Creatinine clearance at least 60 mL/min

Cardiovascular:

* Left ventricular ejection fraction greater than 45%

Pulmonary:

* DLCO greater than 60% of predicted

Other:

* HIV negative
* No active infection
* No concurrent medical condition that would preclude therapy
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks since prior nitrosoureas or mitomycin)

Endocrine therapy:

* Not specified

Radiotherapy:

* No radiotherapy to greater than 30% of bone marrow
* No wide field radiotherapy

Surgery:

* Recovered from any prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-10; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States